CLINICAL TRIAL: NCT06489626
Title: The Effect of a Methylprednisolone Taper on Outcomes Following Total Knee Arthroplasty
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: withdrawn
Sponsor: F. Johannes Plate (Other)
Responsible Party: Sponsor-Investigator, F. Johannes Plate, Director of Research Division of Adult Reconstruction, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY24010173
Record Dates: First submitted 2024-06-28; First posted 2024-07-08 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Arthritis Knee; Knee Osteoarthritis; Pain, Postoperative
Keywords: total knee arthroplasty; knee osteoarthritis; pain management
MeSH Terms: conditions — Osteoarthritis, Knee; Pain, Postoperative; Agnosia | interventions — Calcium Dobesilate

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intraoperative and Post-operative steroid (Experimental): Patients in this groups will receive intraoperative intravenous dexamethasone as well as a 6-day post-operative methylprednisolone taper
  Interventions: Drug: Methylprednisolone 4 milligram Tab; Drug: Dexamethasone injection
- Intraoperative Steroid (Active Comparator): Patients randomized to this group will only receive intraoperative intravenous dexamethasone
  Interventions: Drug: Dexamethasone injection

INTERVENTIONS:
Drug: Methylprednisolone 4 milligram Tab — 6-day 4 milligram methylprednisolone oral taper
  Arms: Intraoperative and Post-operative steroid
Drug: Dexamethasone injection — 4 milligram intravenous dexamethasone will be administered intraoperatively

SUMMARY:
Pain control and early range of motion following total knee arthroplasty are essential for patient satisfaction. Intraoperative steroids (dexamethasone) have been shown to have a significant effect in controlling acute pain following total knee arthroplasty. This study aims to evaluate the effect of a post-operative steroid (methylprednisolone) taper in improving functional and patient-reported outcomes following total knee arthroplasty. A taper means taking a high dose of a medication followed by taking lower doses and each following day until the medication is stopped.

ELIGIBILITY:
Inclusion Criteria:

* Patients indicated for primary total knee arthroplasty.
* Access to computer or smartphone for completion of REDCap surveys

Exclusion Criteria:

* Patients less than 18 years of age, patients unable to consent, known diabetic patients and those with an HgbA1c >6.5 preoperatively, patients who are on chronic steroid treatments, patients with chronic pain on opioid management, patients with allergies to steroids, patients with a history of peptic ulcer disease, patients with a history of heart failure and patients with a history of renal and/or hepatic failure will be excluded. Those that are immunosuppressed as well as pregnant and/or lactating will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Daily Pain at rest and with movement | daily for two weeks
  numeric rating scale from 0 to 10 (0=minimal, 10=maximal) will be used to capture patient experienced pain
Prescription narcotic usage | daily for two weeks
  Oral morphine equivalent units will be collected based on patient usage of prescribed narcotic pain medication
Sleep disturbance | daily for two weeks
  Patients will be asked if pain caused them to be awoken in the night and if so what level of pain they were experiencing at that time
Knee Range of motion | 2-week, 6-week and 3-month postoperative visits
  goniometric measurement of knee extension and flexion

SECONDARY OUTCOMES:
Wound healing | 2-week, 6-week and 3-month postoperative visits
  Surgical site will be evaluated for normal wound healing
Knee Injury and Osteoarthritis Outcome Scores | 2-week, 6-week and 3-month postoperative visits
  Questionnaire assessing for function will be administered (0= extreme problems present, 100= no problems present)

OTHER OUTCOMES:
Postoperative complications | To occur at 30 and 90 days postoperatively
  All complications related to the patients procedure including infection, need for revision, emergency room visits, readmissions, etc. will be collected

CONTACTS AND LOCATIONS:
Overall Officials: Johannes F Plate, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - UPMC East, Monroeville, Pennsylvania
  - UPMC Shadyside Hospital, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wagner ER, Hussain ZB, Karzon AL, Cooke HL, Toston RJ, Hurt JT, Dawes AM, Gottschalk MB. Methylprednisolone taper is an effective addition to multimodal pain regimens after total shoulder arthroplasty: results of a randomized controlled trial: 2022 Neer Award winner. J Shoulder Elbow Surg. 2024 May;33(5):985-993. doi: 10.1016/j.jse.2023.12.016. Epub 2024 Feb 4. PMID 38316236
- [Background] Gottschalk MB, Dawes A, Hurt J, Spencer C, Campbell C, Toston R, Farley K, Daly C, Wagner ER. A Prospective Randomized Controlled Trial of Methylprednisolone for Postoperative Pain Management of Surgically Treated Distal Radius Fractures. J Hand Surg Am. 2022 Sep;47(9):866-873. doi: 10.1016/j.jhsa.2022.06.008. PMID 36058564